CLINICAL TRIAL: NCT06125262
Title: Trajectory Analysis of Neutrophil to Lymphocyte Ratio（NLR） and Its Association With Efficacy of Immunochemotherapy in Esophageal Squamous Cell Carcinoma: A Retrospective Cohort Study
Brief Title: Trajectory Analysis of NLR and Its Association With Efficacy of Immunochemotherapy in ESCC.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, GuiBin Qiao, Professor of Medicine, Guangdong Provincial People's Hospital
Other Study IDs: RICE-Circulation
Record Dates: First submitted 2023-11-05; First posted 2023-11-09 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Esophageal Squamous Cell Carcinoma; Immunotherapy; Chemotherapy
Keywords: Advanced Esophageal Carcinoma; Immunochemotherapy; Trajectory analysis; Blood cell counts
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood cell counts recorded at baseline and after the first cycle of treatment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Conduct a retrospective and prospective study to confirm the association between blood cells counts and the efficacy and safety in immunochemotherapy in patients with advanced esophageal cancer.

DETAILED DESCRIPTION:
Studies have already demonstrated the feasibility of prognostic role of protein biomarkers change during the treatment trajectory of patients in several carcinoma,However, no study focused on the value of trajectory analysis of blood cells counts of Immunochemotherapy in patients with advanced esophageal cancer.

The investigators plan to analyze the dynamic change of blood cells counts longitudinally from preoperation to long term follow-up in advanced esophageal cancer and predict the efficacy and safety of immunochemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed esophageal squamous cell carcinoma
* Potentially resectable esophageal squamous cell carcinoma at first diagnosis (cT1-4a N1-2 M0, cT3-T4a N0M0)
* Treatment-naive
* Expected life span > 6 months
* Aged 18 - 75 years old
* Adequate organ functions
* Performance Status (PS) 0-2
* Participants are fully informed about the whole study and are willing to sign the informed consent

Exclusion Criteria:

* Previous history of thoracic surgery or radiation
* Cervical or multi-origin esophageal cancer
* Known or suspected experimental drug allergy
* Pregnant or lactating women
* Esophagomediastinal fistula
* Peripheral neuropathy
* Previous cancer history other than esophageal cancer
* Severe organ function deterioration that can not tolerate neoadjuvant therapy
* Previous autoimmune diseases
* diabetic history > 10 years
* interstitial pulmonary disease, non-infectious pulmonitis
* Active type B hepatitis
* Any other conditions that may affect patients' safety and compliance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent neoadjuvant immunochemotherapy at Guangdong provincial peoples hospital and The First Affiliated Hospital of Shantou University.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival and disease-free survival. | From the date of diagnosis to the date of death, assessed up to 100 months
  Overall survival rate

SECONDARY OUTCOMES:
Pathologic complete response rate | Three to five working days after surgery
  The rate of pathologic complete response rate after the combined treatment of chemotherapy and immunotherapy following surgery
Objective Response Rate (ORR) | Up to 24 weeks
  Immune-modified Response Evaluation Criteria In SolidTumors (iRECIST) criteria defined complete response and partial response
Major pathological response | Three to five working days after surgery
  ess than 10% residual viable tumor follow neoadjuvant therapy
Event-free survival | From the date of treatment initiation to the date of first progression (local recurrence of tumor or distant metastasis) or death from any cause, assessed up to 100 months
  Event-free survival (EFS)

CONTACTS AND LOCATIONS:
Overall Officials: guibin Qiao, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China